CLINICAL TRIAL: NCT03433547
Title: A Randomized, Open Label, Single Center Study Comparing the Efficacy of Macular Buckle Versus Vitrectomy on Full-thickness Macular Hole and Concurrent Macular Detachment in Eyes With Highly Myopia
Brief Title: Effects of Macular Buckle Versus Vitrectomy on Macular Hole and Macular Detachment in Highly Myopic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Lu, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013meky013-3
Record Dates: First submitted 2018-01-23; First posted 2018-02-14 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Macular Holes; High Myopia; Macular Detachment
Keywords: macular buckling; full-thickness macular hole; macular detachment; internal limiting membrane peeling; high myopia
MeSH Terms: conditions — Retinal Perforations | interventions — Vitrectomy; Gases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buckle (Experimental): Macular buckling, Limbal paracentesis, and intraocular gas injection.
  Interventions: Procedure: Buckle; Other: Limbal paracentesis; Other: Gas injection
- Vitrectomy (Active Comparator): Vitrectomy, peeling internal limiting membrane, and gas tamponade.
  Interventions: Procedure: Vitrectomy; Other: Peeling internal limiting membrane; Other: Gas tamponade

INTERVENTIONS:
Procedure: Buckle — Surgical procedures of macular buckling
  Other Names: Implantation of a device of macular buckling
  Arms: Buckle
Procedure: Vitrectomy — Surgical procedures of small gauge vitrectomy
  Arms: Vitrectomy
Other: Limbal paracentesis — Drainage of aqueous fluid (0.1-0.2 ml) through limbal paracentesis
  Arms: Buckle
Other: Gas injection — Inject gas ( C3F8 100%, 0.2ml-0.3ml) into vitreous cavity through pars plana.
  Arms: Buckle
Other: Peeling internal limiting membrane — Peeling internal limiting membrane with forceps
  Arms: Vitrectomy
Other: Gas tamponade — Filling the vitreous cavity with gas (C3F8, 14%)
  Arms: Vitrectomy

SUMMARY:
Full-thickness macular Hole associated with macular detachment is a one of the maculopathies of high myopia. There is controversy in the primary treatment for this situation. This study will compare the effects of macular buckling versus vitrectomy in a cohort of highly myopic eyes with this situation.

DETAILED DESCRIPTION:
A randomized, open label, single center study comparing the efficacy of macular muckle + gas injection versus internal limiting membrane peeling + gas tamponade on full-thickness macular hole associated with macular detachment in eyes with high myopia.

ELIGIBILITY:
Inclusion Criteria:

* axial length ≥ 26.5 mm or refractive error (spherical equivalent) ≥ 8.0 diopter
* full-thickness macular hole
* macular retinal detachment
* evidence of posterior staphyloma on clinical examination

Exclusion Criteria:

* macular detachment which extended to the peripheral retina (i.e., extension beyond the major vascular arcades in more than one quadrant)
* a history of vitrectomy or scleral buckling
* intraocular active hemorrhage or inflammation
* any media opacity which precluded imaging or clinical evaluation of the macula

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Retinal re-attachment rate | 1 month
  Successful rate of reattachment of macular retina after surgery

SECONDARY OUTCOMES:
Macular hole status | 3 month
  Closure rate of macular hole after surgery on optical coherence tomography
Post-operative best corrected visual acuity | 3 month
  Best corrected visual acuity of the eyes after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lin Lu, MD，PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao X, Li Y, Ma W, Lian P, Yu X, Chen S, Huang X, Liu B, Lu L. Macular buckling versus vitrectomy on macular hole associated macular detachment in eyes with high myopia: a randomised trial. Br J Ophthalmol. 2022 Apr;106(4):582-586. doi: 10.1136/bjophthalmol-2020-317800. Epub 2021 Jan 4. PMID 33397654
- [Derived] Schwartz SG, Flynn HW Jr, Wang X, Kuriyan AE, Abariga SA, Lee WH. Tamponade in surgery for retinal detachment associated with proliferative vitreoretinopathy. Cochrane Database Syst Rev. 2020 May 13;5(5):CD006126. doi: 10.1002/14651858.CD006126.pub4. PMID 32408387